CLINICAL TRIAL: NCT03860324
Title: Erector Spinae vs Fascia Iliaca Block in Hip Arthroplasty Post-operative Analgesia With Erector Spinae Plane Block After Total Hip Replacement Surgery
Brief Title: Erector Spinae vs Fascia Iliaca Block in Hip Arthroplasty
Acronym: ESFIBHA
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Cancelled
Sponsor: Hospital Beatriz Ângelo (Other)
Responsible Party: Principal Investigator, André Carrão, Principal Investigator, Hospital Beatriz Ângelo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 45149
Record Dates: First submitted 2019-02-24; First posted 2019-03-01 (Actual); Last update posted 2021-08-27 (Actual); Status verified 2021-08

CONDITIONS: Pain, Postoperative
Keywords: Hip Arthroplasty; Erector Spinae Plane Block
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control-group (No Intervention): No peripheral nerve block
- Single-shot erector spinae plane block (Experimental): The patient is positioned in lateral decubitus. The anesthesiologist uses a linear high-frequency probe in a longitudinal direction laterally to the mid-sagittal plane at the level of L4 until the transverse process is identified and, more superficial, the erector spinae muscle. A 22G needle of 80mm is introduced in-plane craniocaudally towards the transverse process of L4 until its tip is in the plane deep to the erector spinae muscle. Single-shot block with 30ml of ropivacaine 0,5% + adrenaline 100mcg
  Interventions: Procedure: Single-shot erector spinae plane block
- Single-shot fascia iliaca block (Active Comparator): The patient is positioned in dorsal decubitus. The anesthesiologist uses a linear high-frequency probe in a transversal direction, below the crural arch so as to identify the femoral artery. Afterwards the probe is moved laterally to find the iliac muscle and its fascia. A 22G needle of 80mm is introduced in-plane latero-medially until its tip is below the fascia iliaca (between the muscle and its fascia). Single-shot block with 40ml of ropivacaine 0,2%.
  Interventions: Procedure: Single-shot fascia iliaca block

INTERVENTIONS:
Procedure: Single-shot erector spinae plane block — Single-shot Erector Spinae Plane block with 30ml of ropivacaine 0,5% + adrenaline 150mcg.
  Arms: Single-shot erector spinae plane block
Procedure: Single-shot fascia iliaca block — Single-shot Fascia Iliaca block with 40ml of ropivacaine 0,2%
  Arms: Single-shot fascia iliaca block

SUMMARY:
The thoracic erector spinae plane (ESP) block was first described by Forero et al in September 2016. In their article, the authors presented the possibility of using this block as an option for the control of thoracic neuropathic pain as well as post-operative thoracic pain. The ESP block is done by administering local anesthetic in the plane deep to the erector spinae muscle, which spreads through the costotransverse foramen to the dorsal and ventral roots of the spinal nerves.

Since then, there have been reports about the successful use of this block for bariatric surgery, ventral hernia repair, radical mastectomy, rib fractures, major abdominal surgery and hip replacement. However, there are no studies in the literature comparing the efficacy of the ESP block to other nerve blocks.

The purpose of this study is to compare the post-operative analgesic efficacy of the ESP block to the fascia iliaca (FI) block after total hip replacement (THR).

ELIGIBILITY:
Inclusion Criteria:

* Surgical plan for total hip replacement
* Signing of consent form to participate in the study

Exclusion Criteria:

* Patient refusal
* BMI > 40 kg/m2
* Surgical plan for revision of hip replacement
* Patient unable to quantify pain level
* Chronic kidney disease with a Glomerular Filtration Rate < 50ml/min
* Previously medicated with opioids
* Patient unable to perform the surgery with spinal block
* Allergy to local anesthetics
* Infection in the site of the Erector Spinae Plane or Fascia Iliaca block
* Allergy or contraindication to the use of morphine

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-04-01 (Estimated); Primary Completion 2019-06-30 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Post-operative pain level measured by the Visual Analog Scale | At 6 hours post-operative
  Measurement of patient's pain level using the Visual Analog Scale (with a score of 0-100, 0 being no pain and 100 maximum pain)
Post-operative pain level measured by the Visual Analog Scale | At 12 hours post-operative
  Measurement of patient's pain level using the Visual Analog Scale (with a score of 0-100, 0 being no pain and 100 maximum pain)
Post-operative pain level measured by the Visual Analog Scale | At 24 hours post-operative
  Measurement of patient's pain level using the Visual Analog Scale (with a score of 0-100, 0 being no pain and 100 maximum pain)
Post-operative pain level measured by morphine consumption using patient-controlled intravenous analgesia | At 24 hours post-operative
  Total amount (in mg) of morphine administered by a patient-controlled intravenous analgesia pump of morphine 1mg/ml with bolus of 1ml per patient request with a lockout time of 10 minutes

SECONDARY OUTCOMES:
Muscle Strength grade | At 12 hours post-operative
  Muscle strength grade and comparison with the contralateral limb in the quadriceps femoris muscle
  Muscle strength scale:
  Grade 0: No muscle contraction is detected Grade 1: Muscle contraction is identified but it is insufficient to produce motion Grade 2: The muscle can move the joint only if the force of gravity is eliminated Grade 3: The muscle can move the joint against gravity but without any resistance Grade 4: The muscle can move the joint against moderate resistance Grade 5: The muscle can move the joint against full resistance
Muscle Strength grade | At 24 hours post-operative
  Muscle strength grade and comparison with the contralateral limb in the quadriceps femoris muscle
  Muscle strength scale:
  Grade 0: No muscle contraction is detected Grade 1: Muscle contraction is identified but it is insufficient to produce motion Grade 2: The muscle can move the joint only if the force of gravity is eliminated Grade 3: The muscle can move the joint against gravity but without any resistance Grade 4: The muscle can move the joint against moderate resistance Grade 5: The muscle can move the joint against full resistance
Sensory block assessed through a temperature test | At 24 hours post-operative
  Assessment of sensory block through a temperature test and comparison with the contralateral limb (sensory block vs no sensory block)
Sensory block assessed through a tactile stimulation test | At 24 hours post-operative
  Assessment of sensory block through a tactile stimulation test and comparison with the contralateral limb (sensory block vs no sensory block)
Detection of side effects related to the anesthetic and analgesic technique namely pruritus, urinary retention, nausea and vomiting in each patient | At 24 hours post-operative
  Presence of side effects (pruritus, urinary retention, nausea/vomiting)

CONTACTS AND LOCATIONS:
Overall Officials: André Carrão, Principal Investigator — Hospital Beatriz Ângelo
Locations (1):
- Hospital Beatriz Ângelo, Loures, Lisbon District, Portugal

IPD SHARING:
Plan to Share IPD: No